CLINICAL TRIAL: NCT02581228
Title: Multi-centre, Retrospective, Open Label Study, to Establish and Validate ML-PrediCare for Patients of Advanced Melanoma Undergoing Immunotherapy, as a 1st, 2nd and Later Lines
Brief Title: Multi-Centre, Retrospective, Open Label Study, to Validate ML-PrediCare by Patients With Melanoma Under 1st and 2nd Lines of Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Optimata Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTI-007
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor tissue from an unresectable or metastatic site of disease will be collected for biomarker analyses. Paraffin-embedded tissue samples from patients treated with the immunotherapy drugs (with the previously obtained inform consent form) will be collected from the tissue bank of the hospital and according to the European Commission regulations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Training Set: The objective of the Training stage is to assess the predictive potential of ML-PrediCare for melanoma patients' response to Ipilimumab, Pembrolizumab and Nivolumab.
  Interventions: Device: ML-PrediCare
- Validation Set: The objective of the Validation stage is to test the predictive power of ML -PrediCare in an independent set of patients diagnosed with melanoma.
  Interventions: Device: ML-PrediCare

INTERVENTIONS:
Device: ML-PrediCare

SUMMARY:
This is a retrospective, open label study to establish and validate a prediction technology for advanced melanoma patients under the 1st, 2nd and later treatment lines, with the immunotherapeutic drugs Ipilimumab, Pembrolizumab & Nivolumab, in order to predict response rate and disease progression

DETAILED DESCRIPTION:
The aim of this project is to develop a technology application (termed ML-PrediCare), which is meant to be a predictive stand-alone software device, to support clinicians' decision-making, by predicting the individual patient's response to immunotherapy treatments, e.g., in terms of time-to-progression (TTP).

In Stage I of the study, data will be collected for establishing a training set and assess the predictive potential of the modelling technology for the response of melanoma patients to immunotherapy. In Stage II of the study, data will be collected in order to establish a validation set and test the predictive power of the modelling technology in an independent set of patients diagnosed with melanoma.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for this study:

1. Gender: Female, Male.
2. Age: Eighteen years and older at the start of treatment.
3. Histologically confirmed unresectable Stage III or Stage IV melanoma, as per AJCC staging system.
4. Prior radiotherapy must have been completed at least 2 weeks prior to drug administration.
5. Measurable disease by CT, or PET-CT, or MRI per RECIST 1.1
6. Patient has at least one quantitative measurement of at least one target lesion (primary tumor or metastasis) before treatment.
7. Patient has at least one quantitative measurement of at least one target lesion (primary tumor or metastasis) during or after the treatment.
8. Patient has at least one recorded visit to the treating oncologist before treatment.
9. Patient has at least one recorded visit to the treating oncologist during or after the treatment.
10. Treatment as per SOC for melanoma.

Exclusion Criteria:

Patients meeting one or more of the following criteria are ineligible for this study:

1. History of another malignancy within the previous 2 years except for:

   • Adequately treated Stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 2 years
2. Ocular melanoma
3. Active brain metastases or leptomeningeal metastases.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from up to about 500 melanoma patients will be screened for collection, depending on data availability and completeness of the files
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-04 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint in this study stage is Time to Progression of disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marina Kleiman, PhD, Study Director — Optimata Ltd.; Michal Lotem, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Optimata Ltd., Bne ‘Atarot, Israel

REFERENCES:
- [Derived] Tsur N, Kogan Y, Avizov-Khodak E, Vaeth D, Vogler N, Utikal J, Lotem M, Agur Z. Predicting response to pembrolizumab in metastatic melanoma by a new personalization algorithm. J Transl Med. 2019 Oct 7;17(1):338. doi: 10.1186/s12967-019-2081-2. PMID 31590677